CLINICAL TRIAL: NCT05370690
Title: Retrospective Comparison of the Efficacy of Methotrexate and Azathioprine as Background Treatment for Uveitis of Undetermined Origin: Single-centre Retrospective Study From 2005 to 2020
Acronym: UMetAza
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: UMetAza (29BRC22.0039)
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-02

CONDITIONS: Uveitis
Keywords: Uveitis idiopatic (except anterior), azathioprine, methotrexate
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study at the Brest universitary hospital to evaluate the efficacy of methotrexate (MTX) and azathioprine (AZA) in background treatment of unidentified non anterior uveitis.

DETAILED DESCRIPTION:
Uveitis is a major cause of ocular damage, responsible for 5 to 10% of blindness in the world. More broadly, up to 35% of patients with uveitis have visual acuity impairment ranging from "significant" to "legal blindness" [4]. The figures of "legal blindness" up to 25% according to the studies

The objective of any anti-inflammatory therapy strategy for uveitis is to:

* Quickly control eye inflammation to minimize irreversible structural damage and maintain visual function.
* Prevent inflammatory recurrences, which cause complications and co-morbidity.
* Limit the use of systemic corticosteroids over the course of their deleterious metabolic effects.
* Optimize the risk-benefit balance and promote compliance.

The studies concerning uveitis linked with another disease are multiple and are therefore well documented. Uveitis of undetermined origin is classified, by definition, as uveitis of non-infectious origin.

Anterior uveitis are available for local treatment prior to any discussion of introducing systemic treatment. Intermediate uveitis, posterior and panuveitis justify systemic treatment.

Systemic treatments used in these uveitis are METHOTREXATE, AZATHIOPRINE, MYCOPHENOLATE MOFETIL CICLOSPORINE, INTERFERON ALPHA, anti-TNF alpha. Antimetabolites (azathioprine, mycophenolate mofetil and methotrexate) are the most commonly used immunosuppressants.

Several randomized studies (retrospective or prospective) compared the use of METHOTREXATE (MTX) and MYCOPHENOLATE MOFETIL (MMF), in the management of non-infectious inflammatory ocular disease as a corticosteroid-sparing treatment.

Although MMF has a faster response time compared to MTX for inflammation control, the success rate is equivalent. These studies found no superiority of one molecule over the other .

There are no studies in the literature comparing the use of MTX versus AZA in treatment of these non-prior uveitis of undetermined origin. These two molecules are frequently used in our center as first-line treatment of idiopathic uveitis in an undifferentiated way.

The objective of this study is therefore to determine whether one of these molecules should be preferred for the management of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient age>18 years
* Intermediate, posterior or panuveitis diagnosed clinically by an ophthalmologist.
* Patient treated with azathioprine or methotrexate

Exclusion Criteria:

* Patient under legal protection
* Methotrexate dose < 10mg or azathioprine < 50mg
* Systemic or ophthalmological disease (Behçet, sarcoidosis, Retinopathy of Birdshot, etc.)
* Infectious uveitis
* Ophthalmological surgery < 30 days
* Delayed corticosteroid ocular implant > 3 months
* Introduction of biotherapy simultaneously or prior to immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uveitis (intermediate, posterior or panuveitis) of undetermined origin diagnosed and or followed between January 2005 and March 2020 at the CHRU of Brest and who received treatment with methotrexate or azathioprine.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of methotrexate versus azathioprine in controlling the inflammation of intermediate, posterior and panuveitis of undetermined origin. | one year
  The main evaluation criterion will be the 12-month treatment effectiveness characterized by:
  * No recurrence of inflammation in both eyes as assessed by the patient's referring ophthalmologist
  * Oral corticosteroids <7.5 mg equivalent-prednisone
  * No re-establishment of local corticosteroid therapy > or = at 2 drop/d
  * No treatment stop due to intolerance or adverse reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.